CLINICAL TRIAL: NCT04572854
Title: An Open-Label, Randomized, Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of Pegcetacoplan in the Treatment of Post-Transplant Recurrence of C3G or IC-MPGN
Brief Title: Study Assessing the Safety and Efficacy of Pegcetacoplan in Post-Transplant Recurrence of C3G or IC-MPGN
Acronym: NOBLE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL2-C3G-204
Record Dates: First submitted 2020-09-29; First posted 2020-10-01 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: C3G; IC-MPGN; Renal Transplant; Complement 3 Glomerulopathy; Complement 3 Glomerulopathy (C3G); Dense Deposit Disease (DDD); Membranoproliferative Glomerulonephritis; Membranoproliferative Glomerulonephritis (MPGN); Immune Complex Membranoproliferative Glomerulonephritis (IC-MPGN); C3 Glomerulopathy; C3 Glomerulonephritis; Complement 3 Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Pegcetacoplan treatment of 1080 mg (sub-cutaneous infusion) twice weekly will be given throughout the entire study.
  Interventions: Drug: Pegcetacoplan
- Group 2 (Other): No intervention given during the randomized controlled portion of the study (through week 12). After week 12, subjects will receive pegcetacoplan treatment.
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor

SUMMARY:
This is a Phase 2, multicenter, open-label, randomized, controlled study designed to evaluate the safety and efficacy of pegcetacoplan in patients who have post-transplant recurrence of C3G or IC-MPGN.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at screening
* Must have clinical and pathologic evidence of recurrent C3G or IC-MPGN
* Stable (not improving) or worsening disease, in the opinion of the investigator, in the 2 months preceding the first dose of pegcetacoplan
* eGFR ≥15 mL/min/1.73 m2, calculated by the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) creatinine equation for adults
* No more than 50% glomerulosclerosis or interstitial fibrosis on the screening renal allograft biopsy
* Stable regimen for recurrent C3G/IC-MPGN for at least 4 weeks prior to the screening renal allograft biopsy and from the time of the screening renal allograft biopsy until randomization
* Have received required vaccinations against N. meningitidis, S. pneumoniae, and H. influenzae (type B) or agree to receive vaccinations, if applicable vaccination records are not available. Vaccination is mandatory unless documented evidence exists that subjects are non-responders to vaccination.

Exclusion Criteria:

* Absolute neutrophil count <1000 cells/mm3 during screening
* Previous treatment with pegcetacoplan
* Evidence of rejection on the screening renal allograft biopsy that requires treatment
* Diagnosis or history of HIV, hepatitis B, or hepatitis C infection or positive serology at screening indicative of infection with any of these viruses
* Weight more than 100 kg at screening
* Hypersensitivity to pegcetacoplan or any of the excipients
* History of meningococcal disease
* Malignancy, except for the following:
* Cured basal or squamous cell skin cancer
* Curatively treated in situ disease
* Malignancy free and off treatment for ≥5 years
* Significant renal disease in the renal allograft secondary to another condition (eg, infection, malignancy, monoclonal gammopathy, rejection, or a medication) that would, in the opinion of the investigator, confound interpretation of the study results
* Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedure within 30 days or 5 half-lives from the last dose of the investigational agent (whichever is longer) prior to screening
* Known or suspected hereditary fructose intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (7):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Keck School of Medicine, University of Southern California, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St.Louis, St Louis, Missouri
  - NYU Langone Health Transplant Insitute, New York, New York
  - CUIMC, New York, New York
- Argentina (2):
  - Hospital de Alta Complejidad en Red El Cruce Dr. Nestor Carlos Kirchner, San Juan Bautista, Buenos Aires
  - Hospital Universitario Fundacion Favaloro, Buenos Aires
- Australia (2):
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Monash Medical Centre, Clayton
- Medical University of Vienna, Vienna, Austria
- Brazil (4):
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UPECLIN - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu - FMB/UNESP, Botucatu, São Paulo
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Clinical Research Center, Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- France (3):
  - Lille Regional University Hospital Center, Claude Huriez Hospital, Department of Nephrology, Lille
  - Hopital Edouard Herriot, Hospices Civils de Lyon, Lyon
  - Center Hospitalier Universitaire de Montpellier, Montpellier
- Istituto di Ricerche Farmacologiche Mario Negri IRCCS, Ranica, Italy
- Radbound University Medical Center, Nijmegen, Netherlands
- Hospital Universitario 12 de Octubre, Nephrology Department, Madrid, Spain
- CHUV, Lausanne, Switzerland
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, London
  - Freeman Hospital, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 2, open-label study was conducted in subjects with post-transplant recurrence of complement 3 glomerulopathy (C3G) or immune complex membranoproliferative glomerulonephritis (IC-MPGN) at 23 sites across 11 countries. First subject was recruited on 07 September 2021 and data cut-off (DCO) date was 19 January 2024.
Pre-assignment Details: The study consisted of 2 parts: Part A core study (controlled and non-controlled portion) and Part B long-term extension. A total of 13 subjects were enrolled in the study. Results are presented based on DCO date of 19 January 2024 for Part A. Subjects who experienced clinical benefit from pegcetacoplan administration could participate in part B, a long-term extension, to continue receiving pegcetacoplan until it is commercially available for the disease under study.
Groups:
- Part A: Controlled Portion: Group 1: Subjects received pegcetacoplan 1080 milligram (mg) twice weekly via subcutaneous (SC) infusion on Day 1 and Day 4 of each treatment week until Week 12.
- Part A: Controlled Portion: Group 2: Subjects did not receive any pegcetacoplan treatment until Week 12.
- Part A: Non-controlled Portion: Group 1: Subjects who received pegcetacoplan in Part A controlled portion: Group 1 continued to receive pegcetacoplan 1080 mg twice weekly via SC infusion on Day 1 and Day 4 of each treatment week until Week 52 post Week 12 renal biopsy.
- Part A: Non-controlled Portion: Group 2: Subjects who did not receive pegcetacoplan in Part A controlled portion: Group 2 received pegcetacoplan 1080 mg twice weekly via SC infusion on Day 1 and Day 4 of each treatment week until Week 52 post Week 12 renal biopsy.
Period: Part A: Controlled: Weeks 1 to 12
Arm/Group | Part A: Controlled Portion: Group 1 | Part A: Controlled Portion: Group 2 | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Started | 10 | 3 | 0 | 0
Completed (Subjects completed Part A (controlled portion).) | 10 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part A: Non-controlled: Weeks 13 to 52
Arm/Group | Part A: Controlled Portion: Group 1 | Part A: Controlled Portion: Group 2 | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Started | 0 | 0 | 10 (Subjects rolled over to Part A (non-controlled portion).) | 3 (Subjects rolled over to Part A (non-controlled portion).)
Completed (Subjects completed Part A (non-controlled portion).) | 0 | 0 | 8 | 2
Not Completed | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all subjects who were randomized.
Groups:
- Part A: Controlled Portion: Group 1: Subjects received pegcetacoplan 1080 mg twice weekly via SC infusion on Day 1 and Day 4 of each treatment week until Week 12.
- Total: Total of all reporting groups
Arm/Group | Part A: Controlled Portion: Group 1 | Part A: Controlled Portion: Group 2 | Total
Number analyzed (Participants) | 10 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (12.59) | 44.3 (24.03) | 40.8 (14.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 3 | 12
  Not reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Reduction in C3c Staining on Renal Biopsy at Week 12
Description: C3c staining intensity is semi quantitatively graded on a scale of 0 to 3, in which negative, 1+, 2+ and 3+ staining corresponds to scores of 0 to 3, with 0 being absent and 3 being the highest intensity seen on immunofluorescence. Higher scores indicate worse outcome. Reduction in C3c staining was defined as decrease of at least 2 orders of magnitude of intensity from baseline. Baseline was defined as the most recent non-missing measurement prior to first administration of study drug for Group 1 subjects or randomization for Group 2 subjects.
Time Frame: Baseline (Day 1) and Week 12
Population: The ITT population included all subjects who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: Controlled Portion: Group 1 | Part A: Controlled Portion: Group 2
Number analyzed (Participants) | 10 | 3
Percentage of participants | 50.0 [18.7 to 81.3] | 33.3 [0.8 to 90.6]

2. Secondary Outcome: Percentage of Subjects With Reduction in C3c Staining on Renal Biopsy at Week 52
Description: as for outcome 1
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population included all subjects who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part A: Non-controlled Portion: Group 1: Subjects who received pegcetacoplan in Part A controlled portion: Group 1 continued to receive pegcetacoplan 1080 mg twice weekly via SC infusion on Day 1 and Day 4 of each treatment week until Week 52, post Week 12 renal biopsy.
- Part A: Non-controlled Portion: Group 2: Subjects who did not receive pegcetacoplan in Part A controlled portion: Group 2 received pegcetacoplan 1080 mg twice weekly via SC infusion on Day 1 and Day 4 of each treatment week until Week 52, post Week 12 renal biopsy.
Arm/Group | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Number analyzed (Participants) | 10 | 3
Percentage of participants | 50.0 [18.7 to 81.3] | 66.7 [9.4 to 99.2]

3. Secondary Outcome: Number of Subjects With Shift of C3c Staining From Baseline to Weeks 12 and 52
Description: C3c staining intensity is semi quantitatively graded on a scale of 0 to 3, in which negative, 1+, 2+ and 3+ staining corresponds to scores of 0 to 3, with 0 being absent and 3 being the highest intensity seen on immunofluorescence. Higher scores indicate worse outcome. Baseline was defined as the most recent non-missing measurement prior to first administration of study drug for Group 1 subjects or randomization for Group 2 subjects. Number of subjects who demonstrated a shift of C3c staining from baseline to Week 12 and baseline to Week 52 are presented.
Time Frame: Baseline (Day 1), Week 12 and Week 52
Population: The ITT population included all subjects who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Number analyzed (Participants) | 10 | 3
Participants
  Shift from 3 at baseline to 0 at Week 12 | 3 | 0
  Shift from 2 at baseline to 0 at Week 12 | 1 | 0
  Shift from 3 at baseline to 1 at Week 12 | 1 | 1
  Shift from 2 at baseline to 3 at Week 12 | 0 | 1
  Shift from 3 at baseline to 0 at Week 52 | 4 | 1
  Shift from 2 at baseline to 0 at Week 52 | 0 | 1
  Shift from 3 at baseline to 1 at Week 52 | 1 | 0
  Shift from 2 at baseline to 3 at Week 52 | 1 | 0

4. Secondary Outcome: Percentage of Subjects With Stabilization or Improvement in Estimated Glomerular Filtration Rate (eGFR) at Week 52
Description: eGFR was calculated by using Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) creatinine equation. Stabilization or improvement in eGFR was defined as no more than a 25% decrease relative to baseline. Baseline was defined as the most recent non-missing measurement prior to first administration of study drug for Group 1 subjects or randomization for Group 2 subjects.
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population included all subjects who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Number analyzed (Participants) | 10 | 3
Percentage of participants | 70.0 | 66.7

5. Secondary Outcome: Percentage of Subjects With Stabilization or Improvement of Serum Creatinine Concentration at Week 52
Description: Stabilization or improvement in serum creatinine was defined as no increase or an increase of no more than 25% from baseline. Baseline was defined as the most recent non-missing measurement prior to first administration of study drug for Group 1 subjects or randomization for Group 2 subjects.
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population included all subjects who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Number analyzed (Participants) | 10 | 3
Percentage of participants | 70.0 | 66.7

6. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 52
Description: Blood samples were collected at specified timepoints for analysis of eGFR which was calculated by using CKD-EPI creatinine equation. Baseline was defined as the most recent non-missing measurement prior to first administration of study drug for Group 1 subjects or randomization for Group 2 subjects.
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population included all subjects who were randomized. Only subjects with data collected at baseline and Week 52 are reported.
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73 square meter
Arm/Group | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Number analyzed (Participants) | 9 | 3
milliliter/minute/1.73 square meter | 10.1 (32.67) | -10.3 (14.57)

7. Secondary Outcome: Percentage Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 52
Description: as for outcome 6
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Number analyzed (Participants) | 9 | 3
percentage change | 29.65 (78.707) | -16.67 (21.481)

8. Secondary Outcome: Change From Baseline in Serum Creatinine Concentration at Week 52
Description: Blood samples were collected at specified timepoints for analysis of serum creatinine concentration. Baseline was defined as the most recent non-missing measurement prior to first administration of study drug for Group 1 subjects or randomization for Group 2 subjects.
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Number analyzed (Participants) | 9 | 3
milligram per deciliter | -0.044 (0.8368) | 0.267 (0.4619)

9. Secondary Outcome: Percentage Change From Baseline in Serum Creatinine Concentration at Week 52
Description: as for outcome 8
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
Number analyzed (Participants) | 9 | 3
percentage change | 3.198 (59.5916) | 17.778 (30.7920)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and Treatment-emergent serious adverse events (TESAEs) were collected from first dose of study drug for Group 1 subjects or randomization for Group 2 subjects (Day 1) up to 56 days after the last dose of study drug, approximately 139 days for controlled and 333 days for non-controlled portion. All-cause mortality (deaths) were collected from first dose of study drug (Day 1) up to DCO of 19 January 2024, approximately 864 days.
Description: The safety population included all subjects who received at least 1 dose of pegcetacoplan and subjects who were randomized into Group 2.
Arm/Group | Part A: Controlled Portion: Group 1 | Part A: Controlled Portion: Group 2 | Part A: Non-controlled Portion: Group 1 | Part A: Non-controlled Portion: Group 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/3 | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 5/10 | 0/3 | 5/10 | 0/3
Other Adverse Events (participants affected / at risk) | 7/10 | 3/3 | 8/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Controlled Portion: Group 1 (N=10) | Part A: Controlled Portion: Group 2 (N=3) | Part A: Non-controlled Portion: Group 1 (N=10) | Part A: Non-controlled Portion: Group 2 (N=3)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal tubular disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Controlled Portion: Group 1 (N=10) | Part A: Controlled Portion: Group 2 (N=3) | Part A: Non-controlled Portion: Group 1 (N=10) | Part A: Non-controlled Portion: Group 2 (N=3)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Genital herpes simplex (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyomavirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Loss of bladder sensation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site rash (General disorders) | 1 (23) | 0 (0) | 0 (0) | 0 (0)
Infusion site swelling (General disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
New onset diabetes after transplantation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT04572854/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04572854/SAP_001.pdf